CLINICAL TRIAL: NCT03297931
Title: Comparison of Roasted Pulse Snacks, Pulse Chips and Commercial Snacks on Post-prandial Food Intake, Appetite and Glycemic Response in Healthy Young Adults
Brief Title: Comparison of Pulse Chips and Commercial Snacks on Food Intake, Appetite and Blood Glucose in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SPG_Snack Study
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Diabetes
Keywords: Pulse; Snack; Post-prandial glycemia; Appetite; Food intake; Young adults; Satiety
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Commercial corn chips + Onion dip (Active Comparator): Corn chips + onion dip
  Interventions: Dietary Supplement: Corn Chips + Onion Dip
- Commercial pulse chip + pulse spread (Experimental): Pinto bean chip + hummus
  Interventions: Dietary Supplement: Pinto bean chip + hummus
- Novel pulse chip + pulse spread (Experimental): Yellow pea chip + hummus
  Interventions: Dietary Supplement: Yellow pea chip + hummus
- Commercial pulse chip + non-pulse spread (Experimental): Pinto bean chip + onion dip
  Interventions: Dietary Supplement: Pinto bean chip + onion dip
- Novel pulse chip + non-pulse spread (Experimental): Yellow pea chip + onion dip
  Interventions: Dietary Supplement: Yellow pea chip + onion dip
- Non-pulse chip + pulse spread (Experimental): Corn chips + hummus
  Interventions: Dietary Supplement: Corn chips + hummus

INTERVENTIONS:
Dietary Supplement: Corn Chips + Onion Dip — Non-pulse chip + non-pulse dip
  Arms: Commercial corn chips + Onion dip
Dietary Supplement: Yellow pea chip + hummus — Novel pulse chip + pulse spread
  Arms: Novel pulse chip + pulse spread
Dietary Supplement: Pinto bean chip + hummus — Commercial pulse chip + pulse spread
  Arms: Commercial pulse chip + pulse spread
Dietary Supplement: Pinto bean chip + onion dip — Commercial pulse chip + non-pulse spread
  Arms: Commercial pulse chip + non-pulse spread
Dietary Supplement: Yellow pea chip + onion dip — Novel pulse chip + non-pulse spread
  Arms: Novel pulse chip + non-pulse spread
Dietary Supplement: Corn chips + hummus — Non-pulse chip + pulse spread
  Arms: Non-pulse chip + pulse spread

SUMMARY:
Consumers are often forced to eat fast, convenient foods and snacks ("eat on the go") in order to match the pace of their lifestyles. However, these snack options more often than not offer little health benefit to the consumer. In fact, 55% of calories consumed by Canadians are ultra processed foods, which are limited in their nutrient profile and only offer empty calories. Subsequently, these foods lead the consumer to eat more and provides little to no feelings of satiety or satiation. the proposed objectives of the current project are to examine the physiological benefit(s) of consuming readily available pulse snacks and compare them to other commonly consumed snack varieties. This work aims to incentivize consumers to seek out pulses as valuable snacking options and highlight the benefit of including these as alternatives to other energy-dense snacks that lack the nutritional composition of pulses.

DETAILED DESCRIPTION:
Hypothesis of the study: Inclusion of pulses as part of a snack will lower appetite and post-prandial glycemia (PPG) in comparison to commercial, commonly consumed non-pulse snacks.

Overall Objective of the study: To investigate and compare the effects of pulse and non-pulse snacks served as chips and dip on appetite and PPG in healthy adults.

Specific objectives of the study: To test the acute effects of different pulse snacks on: 1) PPG and appetite for three hours, and 2) food intake 1 hour following consumption of snacks.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and ≤45 years
* BMI: ≥ 18.5 and ≤ 29.9 kg/m2
* Fasting serum glucose: ≤ 5.6 mmol/L
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the Department of Nutritional Sciences. Failure to comply will result in a rescheduled test visit.
* Willing to abstain from alcohol consumption for 24 h prior to all test visits.
* Willing to avoid vigorous physical activity for 24 h prior to all test visits.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Fasting blood glucose > 5.6 mmol/L
* Smoking
* Thyroid problems
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease.
* Presence of gastrointestinal disorder or surgeries within the past year.
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgement.
* Patients who have undergone bariatric surgery at any point.
* Known to be pregnant or lactating.
* Unwillingness or inability to comply with the experimental procedures
* Known intolerance, sensitivity or allergy to pulses or dairy.
* Extreme dietary habits (ie. Atkins diet, very high protein diets, etc.).
* Uncontrolled hypertension (systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg) as defined by the average blood pressure measured at screening.
* Weight gain or loss of at least 10 lbs in previous three months.
* Excessive alcohol intake (more than 2 drinks per day or more than 9 drinks per week)
* Restrained Eaters

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose levels | Starting at the beginning of each session (0 minutes, before consumption of treatment) and every 15 - 30 minutes up to 190 minutes (time of completion of each session)
  Each participant will attend 6 sessions in total (randomized 6-arm cross-over design)
Subjective appetite | Measured every 15-30 minutes up to 190 minutes
  Measured using Visual Analog Scales (VAS)
Food intake | 65 minutes after completion of treatment, 20 minutes is allocated to allow for pizza consumption
  Food intake is measured by the amount of pizza (in grams) consumed during the 20 minute period (pizza is served ad libitum)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey G Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No